CLINICAL TRIAL: NCT03066154
Title: Weekly ModraDoc/r in Combination With Hormonal Treatment and High-dose Intensity-modulated Radiation Therapy in Patients With High-risk Early Stage Prostate Cancer
Brief Title: Oral Docetaxel (ModraDoc/r) in Combination With Hormonal Treatment and Radiation Therapy in High-risk Prostate Cancer
Acronym: DOP
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low inclusion of patients and availability of the IP
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N15DOP
Record Dates: First submitted 2016-09-23; First posted 2017-02-28 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Prostatic Neoplasms
Keywords: High risk prostate cancer; >T2cN+M0
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Ritonavir; Androgen Antagonists; Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- N15DOP (Experimental): Chemoradiation with ModraDoc/r and radiotherapy of the prostate in dose escalation design, followed by maintenance treatment.
  Interventions: Drug: oral docetaxel (ModraDoc/r); Drug: androgen deprivation therapy; Radiation: high-dose intensity-modulated radiation therapy

INTERVENTIONS:
Drug: oral docetaxel (ModraDoc/r) — Weekly once- or twice daily ModraDoc/r
  Other Names: ModraDoc006/ritonavir
Drug: androgen deprivation therapy — ADT according to the standard of care
  Other Names: hormonal therapy
Radiation: high-dose intensity-modulated radiation therapy — 77 Gy in 35 fractions of 2.2 Gy, 5 fractions a week
  Other Names: radiotherapy

SUMMARY:
The optimal treatment for HRPC patients has not yet been established. Recent trials suggest a benefit from early treatment with docetaxel in the castration-sensitive setting, with an improvement in failure free survival in high risk and metastatic patients and increase in overall survival in the metastatic hormone-sensitive group. In these recent randomized controlled trials, patients were treated with hormonal therapy and radiotherapy and adjuvant docetaxel, assuming that early systemic treatment for high risk or metastatic disease could delay progression in patients with aggressive primary tumor characteristics.

With the fact that docetaxel is a known radiosensitizer, combined modality treatment with docetaxel during the radiotherapy could also lead to better local control and reduction of local recurrence. Several phase I and II studies have been done in HRPC patients, to evaluate the combination of high dose radiotherapy and concurrent weekly infusions with docetaxel.

Oral administration of docetaxel has many advantages above intravenously administered drugs for patients. Besides the higher patient convenience, possibly longer treatment duration can be achieved due to better safety. Frequently occurring toxicities of intravenously administered docetaxel, such as neutropenia, hypersensitivity reactions and peripheral polyneuropathy have rarely been observed with the oral docetaxel formulation ModraDoc006/r.

The primary aim of the N15DOP study is to determine the maximum tolerable dose (MTD) of ModraDoc006/r when given in a weekly bidaily schedule in combined modality with high dose intensity radiotherapy and hormonal therapy in castration-sensitive prostate cancer patients with high risk disease, including positive lymph nodes.

DETAILED DESCRIPTION:
Phase IA part This is an open-label, dose-escalating, non-randomized, single centre phase I study of ModraDoc006/r combined with ADT and radiotherapy in patients with high risk prostate cancer, as defined by node positive prostate cancer with all of the following primary tumor characteristics: stage ≥cT2c, Gleason score ≥ 4+3, any PSA level.

Phase IB part After determination of the MTD of ModraDoc006/r in the combined treatment with radiotherapy and hormonal therapy and good tolerability of the treatment without unexpected adverse events during the radiotherapy until 6 weeks after the end of radiotherapy, the study will be further conducted to the phase IB part. This part will explore the feasibility and tolerability of long term treatment with ModraDoc006/r.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven prostate cancer.
2. All eligible patients have hormone naïve non-metastatic node positive high risk prostate cancer. Node positive cancer will be defined as radiological demonstration of more than four pelvic lymph node(s) consisting of bean shaped lymph node(s) with a short axis of minimal 10 mm and/or round lymph node(s) with a minimal size of 8 mm on PSMA, MRI or CT scan.

   PSMA-scans or PET-Choline scans may be used, but are not obligated. Since the use of the PSMA scan is significantly increased in current clinical practice and the chance of false positive results is considered very low in patients with more than 4 positive lymph nodes, histological confirmation of positive lymph nodes is not required for inclusion if more than 4 pathological nodes are seen with the PSMA, MRI or CT scan
3. High risk prostate cancer will be defined as node positive with all of the following primary tumour characteristics: Tumour stage ≥cT2c and Gleason score ≥4+3, any PSA
4. Age ≥ 18 years
5. No signs of metastatic disease on standard diagnostic scans.
6. Normal serum testosterone levels prior to treatment
7. Adequate haematological, renal and hepatic functions

   1. Haemoglobin ≥ 6.0 mmol/l
   2. ANC of ≥ 1.5 x 109 /L
   3. Platelet count of ≥ 100 x 109 /L
   4. Hepatic function as defined by serum bilirubin ≤ 1.5 x ULN, ALAT and ASAT ≤ 2.5 x ULN
   5. Renal function as defined by serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 ml/min (by Cockcroft-Gault formula).
8. WHO performance status of 0-2
9. Able and willing to undergo blood sampling for PK and PD analysis;
10. Life expectancy ≥ 3 months allowing adequate follow up of toxicity evaluation and antitumor activity;
11. Able and willing to swallow oral medication
12. Able and willing to give written informed consent;

Exclusion Criteria:

1. Any treatment with investigational drugs, chemotherapy or immunotherapy within 30 days prior to receiving the first dose of investigational treatment; Patients may be on ADT as long as this is has not been longer than 4 weeks prior the start of the radiotherapy.
2. Patients who have had prior pelvic radiation therapy
3. Patients who have had prior treatment with taxanes
4. TURP within 3 months before start of the study
5. Patients who have had a prostatectomy.
6. Any contra-indication for MRI
7. Major difficulties for marker implantation
8. Unreliable contraceptive methods. Men enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization)
9. Unresolved (> grade 1) toxicities of previous chemotherapy, excluding alopecia.
10. Uncontrolled infectious disease or known Human Immunodeficiency Virus HIV-1 or HIV-2 type patients;
11. Patients with a known history of hepatitis B or C;
12. Bowel obstructions or motility disorders that may influence the resorption of drugs as judged by the treating physician
13. Concomitant use of MDR and CYP3A modulating drugs such as Ca+- entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications, other protease inhibitors, (non) nucleoside analoga, or St. John's wort.
14. Pre-existing neuropathy greater than NCI-CTCAE v4.03 grade 1.
15. Patients with known alcoholism, drug addiction and/or psychiatric of physiological condition which in the opinion of the investigator would impair study compliance; Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.
16. Legal incapacity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose (MTD) of ModraDoc/r in the combination treatment | 12 months
  MTD of ModraDoc006/r (as ModraDoc006 10 mg tablets in combination with one tablet of 100 mg ritonavir) that can safely be administered in a bi-daily weekly schedule in combination with high-dose intensity modulated radiation therapy and androgen-deprivation therapy

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v.4.03 with treatment with ModraDoc006/r in combination with ADT and high dose radiotherapy | 12 months
  Number of participants with treatment-related adverse events as assessed by CTCAE
Number of patients that will have recurrence of prostate cancer after completion of the study treatment | 10 years
  Number of patients that will have recurrence of prostate cancer after completion of the study treatment
Peak Plasma Concentration (Cmax) of docetaxel in this regime. | 12 months
  Peak Plasma Concentration (Cmax) of docetaxel in this regime.
Area under the plasma concentration versus time curve (AUC) of docetaxel in this regime. | 12 months
  Area under the plasma concentration versus time curve (AUC) of docetaxel in this regime.

CONTACTS AND LOCATIONS:
Overall Officials: B van Triest, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vermunt MAC, van der Heijden LT, Hendrikx JJMA, Schinkel AH, de Weger VA, van der Putten E, van Triest B, Bergman AM, Beijnen JH. Pharmacokinetics of docetaxel and ritonavir after oral administration of ModraDoc006/r in patients with prostate cancer versus patients with other advanced solid tumours. Cancer Chemother Pharmacol. 2021 Jun;87(6):855-869. doi: 10.1007/s00280-021-04259-5. Epub 2021 Mar 20. PMID 33744986